CLINICAL TRIAL: NCT04833959
Title: Pilot Study of 89Zr Panitumumab in Pancreas Cancer
Brief Title: Pilot Study of 89-Zr Panitumumab in Pancreas Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-57641; PANC0037 (Other: OnCore); NCI-2021-03447 (Other: CTRP)
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 89Zr-Panitumumab (Experimental): Subjects will be injected with 1 mCi (+/- 20%) of 89Zr-panitumumab followed by PET/CT imaging 4-7 days after study drug injection.
  Interventions: Drug: 89Zr-panitumumab

INTERVENTIONS:
Drug: 89Zr-panitumumab — Imaging Agent

SUMMARY:
The main purpose of the study is to assess the safety of 89Zr-panitumumab as a molecular imaging agent in patients with (metastatic) pancreas cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of pancreatic cancer.

Exclusion Criteria:

* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment.
* History of infusion reactions to monoclonal antibody therapies.
* Pregnant or breastfeeding.
* Subjects receiving Class IA (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents.
* Subjects with a history or evidence of interstitial pneumonitis or pulmonary fibrosis.
* Severe renal disease or anuria.
* Known hypersensitivity to deferoxamine or any of its components.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events assessed by CTCAE v5 | 7 days
  Safety is defined by the number of CTCAE v5 grade 2 or higher adverse events by Day 7 determined that are significant, definitely, probably or possibly related to 89Zr-panitumumab. Safety data will be summarized by grade, severity, and type.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No